CLINICAL TRIAL: NCT05623124
Title: Neurovascular Coupling and Digital Biomarkers in Alzheimer's Disease
Brief Title: Ruijin Neurobank of Alzheimer's Disease and Dementia
Acronym: RJNB-AD
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RJNeuroBank-Dementia
Record Dates: First submitted 2022-10-23; First posted 2022-11-21 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, and DNA extracted from white blood cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dementia: Participants have cognitive impairment and difficulty in daily activity.
  Interventions: Other: No intervention
- Mild cognitive impairment: Participants have cognitive impairment, but no difficulty in daily activity.
  Interventions: Other: No intervention
- cognitively normal: Participants do not have cognitive impairment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to learn about neuroimage and biomarkers in the Alzheimer's continuum. The main questions it aims to answer are:

* How is the neurovascular coupling during AD pathogenesis?
* How is the pattern/mapping of alterations in AD biomarkers? Participants will be observed and visit the research center annually to perform multi-modal MRI, PET, neuropsychological tests, and blood tests.

DETAILED DESCRIPTION:
The observational study recruits participants from clinics and communities with cognitive impairment. Healthy volunteers will also be recruited as controls. Longitudinal observation of these participants will help demonstrate AD biomarkers' significance during AD pathogenesis.

The investigators aim to build an aging population cohort covering the AD continuum and explore key biomarkers for AD. All participants will have multi-modal MRI scanning, PET scanning with different tracers, and blood test. With MRI scanning, the investigators are exploring the effect of neurovascular coupling in AD pathogenesis. In addition, the investigators are trying to find patterns/mapping of AD biomarkers with PET and blood tests. Beyond this, more neuroimage markers and digital biomarkers will be tested in the cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 50 to 90 years old;
2. In accordance with the diagnostic criteria for "mild cognitive impairment due to Alzheimer's disease" and "Dementia" from the National Institutes of Health National Institute on Aging-Alzheimer's Association (NIA-AA) (2011);
3. The Hamilton depression rating scale/17 edition (HAMD) total score<10;
4. The clinical dementia rating (CDR) is 0.5 or above;
5. Neurological examination: no obvious signs;
6. Participants should have a caregiver stable and reliable.
7. Education: primary school (grade 6) or above. They have the ability to complete tests for cognitive ability and have the ability and time to complete regulation of cognitive training

Exclusion Criteria:

1. Other causes of cognitive decline: cerebrovascular disease, central nervous system infection, CJD, Huntington's and Parkinson's disease, DLB, traumatic brain dementia, other physical and chemical factors (such as drugs, alcohol, CO), systemic disease (hepatic encephalopathy, pulmonary encephalopathy, etc.), intracranial occupation (a subdural hematoma, brain tumor), the endocrine system disease (thyroid disease, parathyroid disease), and vitamins deficiency or any other causes of dementia.
2. The history of nervous system diseases, including stroke, optic myelitis, Parkinson's disease, epilepsy, etc.);
3. Psychiatric patients, including schizophrenia or other mental illnesses, bipolar disorder, major depression, or delirium;
4. There are unstable or serious heart, lung, liver, kidney, and hematopoietic system diseases; Poor prognosis because of malignant diseases such as tumors.
5. Vision or hearing problems that lead to poor performance on cognitive tests;
6. Two years history of severe alcoholism, and drug abuse;
7. The researchers believe that the subjects could not complete the study.
8. Contraindication of MRI or PET scanning.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population consists of Alzheimer's disease, mild cognitive impairment, and cognitively normal participants.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
MMSE | once a year
  Mini-mental state examination
Clock drawing test | once a year
  Clock drawing test
Complex figure test | once a year
  Rey-Osterich complex figure test
AVLT | once a year
  Auditory verbal learning test
SDT | once a year
  Symbol-digit test
TMT | once a year
  Trail making test
Naming test | once a year
  Boston naming test
Fluency | once a year
  Language fluency test

SECONDARY OUTCOMES:
Neuroimage markers from MRI | once a year
  Annual changes of volumes of brain
Neuroimage functional markers from fMRI | once a year
  Annual changes of hippocampus related neural connectivity.
Beta-amyloid | once a year
  Annual changes of beta-amyloid in the brain
Tau | once a year
  Annual changes of tau in the brain
SV2A | once a year
  Annual changes of synaptic vesicle 2A in the brain

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
There is not yet a plan to make IPD available to other researchers

REFERENCES:
- [Derived] Xu X, Yang X, Zhang J, Wang Y, Selim M, Zheng Y, Shen R, Sun L, Huang Q, Wang W, Xu W, Guan Y, Liu J, Deng Y, Xie F, Li B; Alzheimer's Disease Neuroimaging Initiative (ADNI). Choroid plexus free-water correlates with glymphatic function in Alzheimer's disease. Alzheimers Dement. 2025 May;21(5):e70239. doi: 10.1002/alz.70239. PMID 40394891